CLINICAL TRIAL: NCT05441657
Title: Visualisation of Changes in Regional Ventilation in Dyspnoeic Postacute COVID-19 Patients: A Case-control Study Using Electrical Impedance Tomography (EIT)
Brief Title: Visualizing Regional Lung Ventilation in Patients With Postacute-COVID-19
Acronym: ViReVentPoCov
Status: Completed | Type: Observational
Sponsor: Jan-Christoph Lewejohann (Other)
Responsible Party: Sponsor-Investigator, Jan-Christoph Lewejohann, Investigator, Jena University Hospital
Organization: Jena University Hospital (Other)
Other Study IDs: KIM-IV-EIT-04
Record Dates: First submitted 2022-06-29; First posted 2022-07-01 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Ventilatory Defect; COVID-19; Post-acute COVID-19 Syndrome; Electric Impedance Tomography; Post-COVID-19 Syndrome
Keywords: post-acute COVID-19 syndrome; EIT; Electric impedance tomographie; long-COVID; post-COVID-19 Syndrome (PCS)
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- dyspnoeic patients with post-acute COVID-19 syndrome: 100 patients with/without persisting dyspnea after COVID-19 disease were examined by Electric Impedance Tomography (EIT).
- control group: 50 healthy volunteers with no lung disease were voluntarily examined by Electric Impedance Tomography.

SUMMARY:
There is a lack of data of spontaneous breathing patients with post-COVID-19 syndrome (PCS) examined by Electrical impedance tomography (EIT). We compare 100 patients with PCS with 50 healthy probands.

DETAILED DESCRIPTION:
When treating patients with dyspnoea, conventional diagnostic tools (computed tomography, spirometry, body plethysmography) often fail to detect pathological changes, making it difficult for the treating physician to choose an appropriate therapeutic approach. Therefore, it would be desirable to have an examination method that reveals the pulmonary changes in postacute Corona-Virus-Disease-2019 (COVID-19) syndrome (PCS) patients that remain hidden from other diagnostic procedures.

Electrical impedance tomography (EIT) is a non-invasive and radiation-free imaging technique that can show the regional ventilation of the lungs almost "in real-time" based on the changes in the electrical impedance of the thorax during inspiration and expiration. This method is based on the observation that the electrical conductivities of biological tissues vary considerably depending on their nature and functional state. Clinical questions in which the inhomogeneity of lung ventilation is to be analysed (e.g., under- or overinflation of individual lung areas, lung collapse, etc.) can be investigated particularly well with EIT since intrathoracic impedance changes correlate strongly with changes in regional lung ventilation.

Up to now, EIT has mainly been used as a monitoring method in intensive care medicine to adapt ventilation settings and other therapeutic measures to the individual needs of patients. In this field, the method has proven useful for obtaining an overview of the distribution of a respiratory volume in a transverse EIT slice, comparing different lung regions, identifying inhomogeneities and assessing regional ventilation during spontaneous breathing.

The aim of this case-control study is to use EIT data obtained during routine examinations of post-COVID patients to analyse whether patients with PCS show more distinct lung alterations than the control group. Maybe these lung alterations correlate with dyspnea most patients report subjectively.

ELIGIBILITY:
Inclusion Criteria:

* for control group: no current lung diseases, over 18 years old
* for patients with postacute COVID-19 syndrome: over 18 years, positive SARS-CoV-2-PCR

Exclusion Criteria:

* heart pacemaker
* epilepsy
* BMI over 50

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 patients with postacute COVID-19 syndrome who present themselves at the outpatient clinic of the University hospital in Jena (JUH) were examined by EIT. 50 lunghealthy volunteers were examined by EIT at JUH.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
pathogenic changes in regional lung ventilation | until July 2022
  pathogenic changes in regional lung ventilation considered

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Christoph Lewejohann, Dr.med., Study Director — Jena University Hospital
Locations (1):
- Jena university hospital, Jena, Thuringia, Germany

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/57/NCT05441657/Prot_SAP_000.pdf